CLINICAL TRIAL: NCT07122635
Title: Effectiveness of Dry Eye Treatment With Diquafosol Sodium 3% After Phaco Surgery
Status: Completed | Type: Observational
Sponsor: Le Xuan Cung (Other)
Responsible Party: Sponsor-Investigator, Le Xuan Cung, Head of Cornea Department, Vietnam National Eye Hospital
Organization: Vietnam National Eye Hospital (Other)
Other Study IDs: 764/QD-BVMTW No. 17
Record Dates: First submitted 2025-07-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye Disease
Keywords: Diquafosol; dry eye; phaco surgery; cataract surgery
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing phacoemulsification surgery and having dry eye 1 week after the surgery
  Interventions: Drug: Diquafosol Sodium 3%

INTERVENTIONS:
Drug: Diquafosol Sodium 3% — Diquafosol Sodium 3% ophthalmic solution, 1 drop each time, 6 times daily, from baseline (1 week after the surgery) to 12 weeks

SUMMARY:
The goal of this observational study is to evaluate the effectiveness of diquafosol sodium 3% in patients undergoing phacoemulsification surgery and having dry eye 1 week after the surgery. The main question it aims to answer is whether using diquafosol will help improve symptoms and signs of dry eye in patients after phaco surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing phacoemulsification surgery with IOL implantation
* Diagnosis with grade 1, grade 2 or grade 3 dry eye one week after the surgery according to DEWS 2007 classification and Sullivan's severity grading scheme

Exclusion Criteria:

* Patients with grade 3 or 4 dry eye before phaco surgery
* Phaco surgery with complications during or after surgery
* Patients with other eye surgeries within 6 months before phaco surgery
* Patients who are using other eye drops before phaco surgery, except artificial tears
* Patients with acute eye infections
* Patients who do not return for follow-up appointments
* Patients who do not comply with treatment
* Patients having allergy with diquafosol 3%
* Patients having side effects with diquafosol 3% and do not want to continue using the drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with grade 1, grade 2 or grade 3 dry eye according to DEWS 2007 classification and Sullivan's severity grading scheme one week after phacoemulsification surgery with IOL implantation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Change in OSDI score | From starting diquafosol (baseline) to 12 weeks
  Change in OSDI score after treatment with diquafosol from baseline (1 week after surgery) to 4 weeks, 8 weeks, 12 weeks.
  At the preoperative and postoperative examinations, patient will be evaluated dry eye symptoms according to the OSDI questionnaire (from 0-100 points)
Change in Tear film breakup time (TBUT) score | From starting diquafosol (baseline) to 12 weeks
  Change in tear film breakup time (TBUT) score after treatment with diquafosol from baseline (1 week after surgery) for 4 weeks, 8 weeks, 12 weeks.
  At the preoperative and postoperative examinations, patient will be evaluated tear film breakup time which is measured after fluorescein staining. At each examination, TBUT score is measured 3 times to calculate the average value.

SECONDARY OUTCOMES:
Change in Schirmer I test value | From starting diquafosol (baseline) to 12 weeks
  Change in Schirmer I test value after treatment with diquafosol from baseline (1 week after surgery) for 4 weeks, 8 weeks, 12 weeks.
  At the preoperative and postoperative examinations, patient will be evaluated total tear secretion using the Schirmer I test.
Change in Tear meniscus height | From starting diquafosol (baseline) to 12 weeks
  Change in Tear meniscus height after treatment with diquafosol from baseline (1 week after surgery) for 4 weeks, 8 weeks, 12 weeks.
  At the preoperative and postoperative examinations, tear meniscus height will be measured using TMH mode on Keratograph 5M machine.
Change in Corneal staining score | From starting diquafosol (baseline) to 12 weeks
  Change in corneal staining score after treatment with diquafosol from baseline (1 week after surgery) for 4 weeks, 8 weeks, 12 weeks.
  At the preoperative and postoperative examinations, patient will be evaluated corneal staining score, which is measured after fluorescein staining and calculated according to NEI grading scale.
Change in Conjunctival staining score | From starting diquafosol (baseline) to 12 weeks
  Change in conjunctival staining score after treatment with diquafosol from baseline (1 week after surgery) for 4 weeks, 8 weeks, 12 weeks.
  At the preoperative and postoperative examinations, patient will be evaluated conjunctival staining score, which is measured after Lissamine green staining and calculated according to NEI grading scale.
Change in Tear film breakup pattern | From starting diquafosol (baseline) to 12 weeks
  Change in tear film breakup pattern from baseline (1 week after surgery) and after 12 weeks of treatment with diquafosol.
  Tear film breakup pattern will be assessed after fluorescein staining.

OTHER OUTCOMES:
Rate of side effects of diquafosol | From starting diquafosol (baseline) to 12 weeks
  Rate of side effects of diquafosol will be assessed at each examination.
Influence of Risk Factors on Treatment Effectiveness | From starting diquafosol (baseline) to 12 weeks
  The influence of risk factors on treatment effectiveness will be evaluated (yes or no, influence or not). A Fisher's Exact Test will determine if there is a statistically significant difference (p<0.05) between subgroups of a specific risk factor.

CONTACTS AND LOCATIONS:
Locations (1):
- Vietnam National Eye Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided